CLINICAL TRIAL: NCT05036850
Title: China Kidney Patient Trials Network
Acronym: CKPTN
Status: Recruiting | Type: Observational
Sponsor: George (Beijing) Clinical Research Co. Ltd. (Industry)
Responsible Party: Sponsor
Organization: Emerald Clinical Inc. (Industry)
Other Study IDs: CKPTN2019
Record Dates: First submitted 2021-08-27; First posted 2021-09-08 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Kidney Diseases
Keywords: Chronic Kidney Disease; Diabetic Nephropathy; Hypertensive Kidney Disease; Glomerulonephritis; GN; Focal Segmental Glomerulosclerosis; FSGS; Membranous Nephropathy; Minimal Change Disease; IgA Nephropathy; Glomerulonephritis not otherwise specified
MeSH Terms: conditions — Kidney Diseases; Renal Insufficiency, Chronic; Diabetic Nephropathies; Hypertensive Nephropathy; Glomerulonephritis; Glomerulosclerosis, Focal Segmental; Glomerulonephritis, Membranous; Nephrosis, Lipoid; Glomerulonephritis, IGA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Incident and Prevalent Patients: Incident and prevalent patients diagnosed with a kidney disease at participating centres

SUMMARY:
This is a prospective multi-centre, observational cohort study of incident and prevalent patients diagnosed with a kidney disease in China.

ELIGIBILITY:
Inclusion Criteria:

1. Documented diagnosis of primary kidney disease
2. Regular visits (at least 6 monthly) with a physician at a participating site
3. eGFR > 15 ml/min/1.73 m2
4. ≥ 2 years of age
5. Willing and able to sign informed consent
6. Willing to be approached about participation in interventional research studies

Exclusion Criteria:

* 1. Life-expectancy of less than 6 months

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be recruited from units that provide a comprehensive nephrology service
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2021-09-27 (Actual); Primary Completion 2026-09-15 (Estimated); Study Completion 2031-02-28 (Estimated)

PRIMARY OUTCOMES:
eGFR (estimated Glomerular Filtration Rate) | Collected six monthly, up to 5 years
  Routine results
Albuminuria | Collected six monthly, up to 5 years
  Routine results

CONTACTS AND LOCATIONS:
Locations (1):
- George Clinical (Beijing), Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The current plan is that only aggregate data will be shared for research purposes. IPD would only be reviewed in incidental findings and only be discussed with the participant in question.

REFERENCES:
- [Background] Luyckx VA, Tonelli M, Stanifer JW. The global burden of kidney disease and the sustainable development goals. Bull World Health Organ. 2018 Jun 1;96(6):414-422D. doi: 10.2471/BLT.17.206441. Epub 2018 Apr 20. PMID 29904224
- [Background] Tonelli M, Muntner P, Lloyd A, Manns BJ, Klarenbach S, Pannu N, James MT, Hemmelgarn BR; Alberta Kidney Disease Network. Risk of coronary events in people with chronic kidney disease compared with those with diabetes: a population-level cohort study. Lancet. 2012 Sep 1;380(9844):807-14. doi: 10.1016/S0140-6736(12)60572-8. Epub 2012 Jun 19. PMID 22717317
- [Background] Go AS, Chertow GM, Fan D, McCulloch CE, Hsu CY. Chronic kidney disease and the risks of death, cardiovascular events, and hospitalization. N Engl J Med. 2004 Sep 23;351(13):1296-305. doi: 10.1056/NEJMoa041031. PMID 15385656
- [Background] McGrogan A, Franssen CF, de Vries CS. The incidence of primary glomerulonephritis worldwide: a systematic review of the literature. Nephrol Dial Transplant. 2011 Feb;26(2):414-30. doi: 10.1093/ndt/gfq665. Epub 2010 Nov 10. PMID 21068142
- [Background] Strippoli GF, Craig JC, Schena FP. The number, quality, and coverage of randomized controlled trials in nephrology. J Am Soc Nephrol. 2004 Feb;15(2):411-9. doi: 10.1097/01.asn.0000100125.21491.46. PMID 14747388
- [Background] Perkovic V, Craig JC, Chailimpamontree W, Fox CS, Garcia-Garcia G, Benghanem Gharbi M, Jardine MJ, Okpechi IG, Pannu N, Stengel B, Tuttle KR, Uhlig K, Levey AS. Action plan for optimizing the design of clinical trials in chronic kidney disease. Kidney Int Suppl (2011). 2017 Oct;7(2):138-144. doi: 10.1016/j.kisu.2017.07.009. Epub 2017 Sep 20. PMID 30675428
- [Background] de Zeeuw D, Heerspink HJL, Jardine M, Perkovic V. Renal trials in diabetes need a platform: time for a global approach? Lancet Diabetes Endocrinol. 2018 May;6(5):356-358. doi: 10.1016/S2213-8587(17)30263-2. Epub 2017 Aug 7. No abstract available. PMID 28797748